CLINICAL TRIAL: NCT03396601
Title: Administration of Intravenous NRX100 (Ketamine) vs Placebo Infusion for Rapid Stabilization of Acute Suicidal Ideation and Behavior in Patients With Bipolar Depression
Brief Title: NRX100 vs. Placebo for Rapid Stabilization of Acute Suicidal Ideation and Behavior in Bipolar Depression
Acronym: SevereBD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NeuroRx, Inc. (Industry)
Collaborators: Target Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NRX100_001
Record Dates: First submitted 2018-01-05; First posted 2018-01-11 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Bipolar Depression; Suicidal Ideation
MeSH Terms: conditions — Bipolar Disorder; Suicidal Ideation | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and Care Providers will be masked with regard to medication administered. Outcomes Assessors will not be present during IV infusion of medication.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NRX-100 infusion (Experimental): Infusion of IV NRX-100 (ketamine)
  Interventions: Drug: Ketamine Hydrochloride
- Saline (placebo) infusion (Experimental): Infusion of IV Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Ketamine HCl will be infused intravenously at a dose of 0.5 mg/kg over 40 minutes
  Arms: NRX-100 infusion
Drug: Placebo — Normal Saline placebo will be infused IV over 40 minutes
  Arms: Saline (placebo) infusion

SUMMARY:
NMDA antagonist drugs have increasingly been demonstrated to reduce symptoms of depression and suicidal ideation. NeuroRx has developed a sequential therapy consisting of IV NRX-100 (ketamine HCL) for rapid stabilization of symptoms of depression and suicidal ideation followed by oral NRX-101 (fixed dose combination of D-cycloserine and lurasidone) for maintenance of stabilization from symptoms of depression and suicidal ideation. This study will test the hypothesis that that NRX-100 is superior to placebo in achieving rapid reduction in symptoms of depression and suicidal ideation in patients with Severe Bipolar Depression and Acute Suicidal Ideation or Behavior within 24 hours of administration.

DETAILED DESCRIPTION:
Background and Rationale: NMDA antagonist drugs have increasingly been demonstrated to reduce symptoms of depression and suicidal ideation. Specifically, NRX-100 (ketamine HCl, 0.5 mg/kg IV over 40 minutes) has been shown to induce acute reductions in suicidality and depression in patients with bipolar depression, relative to control. Numerous reports have documented a 50% reduction in the MADRS depression scale and a 75% reduction in suicidality following a single infusion of ketamine in patients with suicidal ideation and depression. While the repeat use of ketamine is not supported and may be contraindicated by the literature, D-cycloserine (DCS), when combined with SSRI antidepressants in patients with treatment resistant depression, and when combined with atypical antipsychotics, in particular lurasidone (NRX-101), has shown separation from control and ability to maintain remission from suicidality and depression over 6 weeks with oral use.

Primary Objective:

• To test the hypothesis that a single infusion of NRX-100 is superior to placebo infusion in the rapid stabilization of patients with severe Bipolar Depression and Acute Suicidal Ideation and Behavior (ASIB).

Secondary Objectives:

• Key secondary: To test the hypothesis that there is a more favorable reduction in the mean change from baseline on the Montgomery Asberg Depression Rating Scale (MADRS) between NRX-100 and saline groups on day 1 and day 2.

Methodology: A multi-center, randomized, double-blind, trial involving a single IV infusion to achieve response by 24 hours. The randomization will be 3:1 favoring NRX-100 (ketamine) infusion (n=105) vs. Saline infusion (n=35). Subjects who respond successfully to treatment will be offered enrollment in a six week followup study of NRX-101 (an oral fixed dose combination of d-cycloserine and lurasidone) vs. standard of care in order to ascertain maintenance of the ketamine effect.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. 18 to 65 years of age, inclusive, at screening.
2. Able to understand and provide written and dated informed consent prior to screening. Deemed likely to comply with study protocol and communicate AEs and other clinically important information, and agree to be hospitalized to complete screening and initiate experimental treatment.
3. Resides in a stable living situation, in the opinion of the investigator
4. Has an identified reliable informant, in the opinion of the investigator
5. Diagnosed with bipolar disorder (BD) according to the criteria defined in the DSM-5. The diagnosis of BD will be made by a psychiatrist and supported by the MINI 7.0.2.
6. Suicidal ideation or behavior as evidenced by an answer of "Yes" to item 4 or item 5 on the C-SSRS.
7. A score of greater than or equal to 20 on the 10 items of the BISS that correspond with MADRS (equivalent to MADRS (BDM) total score of 30).
8. In good general health, as ascertained by medical history, physical examination (including measurement of seated vital signs), clinical laboratory evaluations, and electrocardiogram
9. If female, a status of non-childbearing potential or use of an acceptable form of birth control per the following specific criteria:

   1. Non-childbearing potential (e.g., physiologically incapable of becoming pregnant, i.e., permanently sterilized [status post hysterectomy, bilateral tubal ligation], or post-menopausal with last menses at least one year prior to screening); or
   2. Childbearing potential, and meets the following criteria:

   i. Using any form of hormonal birth control, on hormone replacement therapy started prior to 12 months of amenorrhea, using an intrauterine device (IUD), having a monogamous relationship with a partner who has had a vasectomy, or sexually abstinent.

   ii. Negative urinary pregnancy test at screening, confirmed by a second negative urinary pregnancy test at randomization prior to receiving study treatment.

   iii. Willing and able to continuously use one of the following methods of birth control during the course of the study, defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly: implants, injectable or patch hormonal contraception, oral contraceptives, IUD, double-barrier contraception, sexual abstinence. The form of birth control will be documented at screening and pre-ketamine baseline.
10. Body mass index between 18-35kg/m2.
11. Concurrent psychotherapy will be allowed if the type and frequency of the therapy (e.g., weekly or monthly) has been stable for at least three months prior to screening and is expected to remain stable for the duration of the study.
12. Concurrent hypnotic therapy (e.g., with zolpidem, zaleplon, melatonin, benzodiazepines, or trazodone) will be allowed if the therapy has been stable for at least four weeks prior to screening and if it is expected to remain stable during the course of the subject's participation in the study. Subjects can also continue treatment with benzodiazepines used for anxiety if therapy has been stable for at least four weeks prior to screening and if it is expected to remain stable during the course of the subject's participation in the study.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study.
2. Female who is pregnant or breastfeeding.
3. Female with a positive pregnancy test at screening or before oral dosing of investigational product.
4. Current DSM-5 diagnosis of moderate or severe substance use disorder (except marijuana or tobacco use disorder) within the 12 months prior to screening. Substance abuse cannot be the precipitant of entry to treatment.
5. Subjects with a lifetime history of PCP/ketamine drug use, or failed use of ketamine for depression.
6. History of schizophrenia or schizoaffective disorder, or any history of psychotic symptoms when not in an acute bipolar mood episode.
7. History of anorexia nervosa, bulimia nervosa, or eating disorder NOS (OSFED) within five years of screening.
8. Has dementia, delirium, amnestic, or any other cognitive disorder.
9. Any major psychiatric disorder, including a personality disorder, which is clinically predominant to BD at screening, or has been the primary focus of treatment predominant to BD at any time within six months prior to screening.
10. Current major psychiatric disorder, diagnosed at screening with the MINI 7.0.2, that is the primary focus of treatment, with BD as the secondary focus of treatment, within the past six months.
11. A clinically significant abnormality on the screening physical examination that might affect safety or study participation, or that might confound interpretation of study results according to the study clinician.
12. Current episode of:

    1. Untreated hypertension, (Stage 1 or greater) as defined by a systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg at screening on two of three measurements at least 15 minutes apart. If untreated due to missing medication dose/s this is not exclusionary.
    2. Hypertension, Stage 2, as defined by a systolic blood pressure ≥155 mmHg or diastolic blood pressure ≥99 mmHg within 1.5 hours prior to ketamine infusion on two of three measurements at least 15 minutes apart at the pre-ketamine assessment (on Day 0 at Visit 1).
    3. Recent myocardial infarction (within one year).
    4. Syncopal event within the past year.
    5. Congestive heart failure (CHF) New York Heart Association Criteria >Stage 2.
    6. Angina pectoris.
    7. Heart rate <50 or >105 beats per minute at screening, pre-ketamine infusion (Day 0) or at randomization (Day 1).
    8. QTcF ≥450 msec at screening for men, ≥ 470 msec for women, pre-ketamine infusion (Day 0), or at randomization (Day 1), on two of three measurements at least 15 minutes apart.
13. History of hypertension, or on antihypertensives for the purpose of lowering blood pressure, with either an increase in antihypertensive dose or increase in the number of antihypertensive drugs used to treat hypertension over the last two months.
14. Chronic lung disease, excluding asthma.
15. Lifetime history of surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system (CNS) disorder (e.g., Alzheimer's or Parkinson's Disease), epilepsy, mental retardation, or any other disease/procedure/accident/intervention that, according to the screening clinician, is deemed associated with significant injury to or malfunction of the CNS; or history of significant head trauma within the past two years.
16. Presents with any of the following lab abnormalities:

    a. Subjects with diabetes mellitus fulfilling any of the following criteria: i. Unstable diabetes mellitus defined as glycosylated hemoglobin (HbA1c) >8.0 % at screening.

    ii. Admitted to hospital for treatment of diabetes mellitus or diabetes mellitus-related illness in the past 12 weeks.

    iii. Not under physician care for diabetes mellitus. iv. Has not been on the same dose of oral hypoglycemic drug(s) and/or diet for the four weeks prior to screening. For thiazolidinediones (glitazones) this period should not be less than eight weeks.

    b. Any other clinically significant abnormal laboratory result (as determined by the investigator and medical monitor) at the time of the screening.
17. Any current or past history of any physical condition which, in the investigator's opinion, might put the subject at risk or interfere with study results interpretation.
18. Subjects on exclusionary concomitant psychotropic medications (see Appendix 1) as defined in the study manual.
19. At randomization, subjects prescribed more than one agent in each category;

    1. Approved antidepressants (e.g., SSRIs, SNRIs, TeCAs, fluoxetine), but not 5-HT-2a antagonists (lurasidone, aripiprazole, olanzapine, quetiapine)
    2. Mood stabilizers (e.g., lithium, carbamazepine, valproic acid)
20. Subjects with exclusionary laboratory values (see Table 2).
21. Known allergies to lurasidone or Latuda, cycloserine or Seromycin, or the excipients mannitol, croscarmellose sodium, magnesium stearate, silicon dioxide, and/or HPMC (hydroxypropylmethylcellulose).
22. Participation in any clinical trial with an investigational drug or device within the past month or concurrent to study participation.
23. Study site personnel and/or persons employed by NeuroRx, Inc. or Target Health or by the investigator or study site (i.e., permanent, temporary contract worker, or designee responsible for the conduct of the study), or an immediate family member (i.e., spouse or parent, child, or sibling [biological or legally adopted]) of such persons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Suicidal Ideation | 24 hours
  A score of 3 or less on the Columbia Suicidality Severity Rating Scale (C-SSRS). The scale is scored from 0 to 5 on suicidal ideation.

SECONDARY OUTCOMES:
Depression | 24 hours
  Mean change from baseline on Montgomery Asberg Depression Rating Scale (MADRS) between NRX-100 and saline infusion. The scale consists of 10 items, each scored from 0-6, for a possible total score of 60.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Brecher, MD, Study Director — VP, Clinical Development, NeuroRx, Inc.
Locations (2):
- United States (2):
  - Research Centers of America, Hollywood, Florida
  - JP Smith Hospital, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No